CLINICAL TRIAL: NCT06175351
Title: A Randomized, Double-Blind, Placebo-Controlled Phase Ib/IIa Clinical Study to Evaluate the Pharmacokinetic Characteristics, Safety, Tolerability, and Preliminary Efficacy of 9MW1911 in Patients With Moderate to Severe Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: Study to Evaluate the Pharmacokinetic Characteristics, Safety, Tolerability, and Preliminary Efficacy of 9MW1911 in Patients With Chronic Obstructive Pulmonary Disease (COPD).
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Mabwell (Shanghai) Bioscience Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 9MW1911-2022-CP103
Record Dates: First submitted 2023-12-04; First posted 2023-12-18 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-05

CONDITIONS: Moderate to Severe Chronic Obstructive Pulmonary Disease (COPD)

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Phase Ib 9MW1911 (Experimental): 9MW1911 is administered intravenously in a multiple ascending dose pattern in four dose levels. Each level includes 6 patients.
  Interventions: Drug: 9MW1911
- Phase IIa 9MW1911 (Experimental): 9MW1911 is administered intravenously (two doses selected on phase Ib). Each dose level includes up to 18 patients.
  Interventions: Drug: 9MW1911
- Phase Ib Placebo (Placebo Comparator): Placebo is administered intravenously in a multiple ascending dose pattern in four dose levels. Each level includes 2 patients.
  Interventions: Drug: Placebo
- Phase IIa Placebo (Placebo Comparator): Placebo is administered intravenously (two doses selected on phase Ib). Each dose level includes up to 6 patients.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: 9MW1911 — Participants will receive IV 9MW1911 every 4 weeks.
  Arms: Phase IIa 9MW1911; Phase Ib 9MW1911
Drug: Placebo — Participants will receive IV placebo every 4 weeks.
  Arms: Phase IIa Placebo; Phase Ib Placebo

SUMMARY:
The study will evaluate the pharmacokinetic characteristics, safety, tolerability, and preliminary efficacy of 9MW1911 in combination with standard of care COPD maintenance therapy in patients with moderate to severe COPD.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients must be >=40 years of age and capable of giving signed informed consent.
2. Body Mass Index (BMI) of 16 kg/m² to 32 kg/m².
3. Documented physician diagnosis of COPD for at least 1 year.
4. Smoking history with a minimum of 10 pack-year.
5. Post-bronchodilator of FEV1>=30 and <80% of predicted normal value at screening.
6. Modified Medical Research Council (dyspnea scale) (mMRC) score>=2.
7. COPD assessment score (CAT) score >=10, with each of the phlegm and cough items with a score >=2.
8. Documented stable, standard-of-care COPD maintenance therapy for at least 8 weeks prior to screening, with no anticipated changes during the screening period and throughout the study.
9. Documented history of >= 2 moderate or >=1 severe COPD exacerbations within 12 months prior to screening.

Exclusion Criteria:

1. Current diagnosis of asthma according to the Global Initiative for Asthma guidelines or other accepted guidelines, or documented history of asthma.
2. Diagnosis of Alpha-1 Antitrypsin Deficiency.
3. Moderate to severe COPD exacerbation, within 4 weeks prior to randomization.
4. History of lung pneumonectomy, or lung volume reduction within 12 months prior to screening.
5. Clinically significant respiratory disease other than COPD that significantly affect the study.
6. Evidence of active injection with Mycobacterium tuberculosis or nontuberculous mycobacteria, latent, or inadequately treated infection with Mycobacterium tuberculosis.
7. COVID-19 vaccination injection within 14 days before randomization.
8. Long-term treatment with oxygen (oxygen therapy time >15h/day), or treatment with mechanical ventilation
9. Clinically significant sleep apnea requiring continuous positive airway pressure (CPAP) or non-invasive positive pressure ventilation (NIPPV).
10. Participating in, or scheduled for a pulmonary rehabilitation program within 4 weeks of screening.
11. Clinically significant abnormal electrocardiogram (ECG) at randomization that may affect the conduct of the study.
12. Myocardial infarction, unstable angina, or stroke occurring within 12 months prior to screening;
13. Heart failure (NYHA Class III or IV) within 6 months prior to screening.
14. Uncontrolled hypertension (ie, systolic blood pressure>180 mmHg or diastolic blood pressure >110 mmHg with or without use of anti-hypertensive therapy).
15. Treatment with other biological agents (including anti-IL4, IL-5, IL-13 monoclonal antibodies) or immunosuppressive therapy within 2 months prior to screening.
16. Alcohol or drug abuse within 1 year prior to screening.
17. Malignancy, current or within the past 5 years. Suspected malignancy or undefined neoplasms.
18. Positive test for Hepatitis B surface antigen (HbsAg), Hepatitis C virus antibody (HCVAb), Syphilis Treponema pallidum antibody (Syphilis TP), or Human Immunodeficiency Virus (HIV Ag/Ab).
19. Alanine aminotransferase (ALT) >= 2 times the upper limit of normal (ULN); Aspartate aminotransferase (AST) >= 2 times ULN; Total bilirubin >= 1.5 times ULN.
20. Estimated glomerular filtration rate (eGFR) <60 mL/min/1.73m2.
21. History of systemic allergic reaction (including systemic allergic reaction to any biological therapy), or history of immediate allergic reaction to any biological therapy.
22. Participation in an interventional clinical studies within 3 months that could affect the result of this study.
23. Pregnant or lactating women. Women of child-bearing potential (WOCBP) with a positive blood serum pregnancy test at screening. Planning a pregnancy during the intervention period and for at least 20 weeks after the last dose of study intervention. Subjects of child-bearing potential (including female subjects, male subjects and their female partners of child-bearing potential) unable to use reliable contraception during the intervention period and for at least 20 weeks after the last dose of study intervention.
24. Confirmed COVID-19 infection at screening. Known history of COVID-19 infection within 4 weeks prior to screening. History of requiring mechanical ventilation or extracorporeal membrane oxygenation (ECMO) secondary to COVID-19 within 3 months prior to screening. Participants who have had a COVID-19 infection prior screening have not yet sufficiently recovered to participate in the procedures of a clinical trial.
25. Life expectancy of no more than 12 months.
26. Subjects who is inappropriate to participate in the trial due to any reasons as determined by the investigator.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-07-06 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Pharmacokinetic characteristics. | 36 weeks
  Peak concentration (Cmax)
Pharmacokinetic characteristics. | 36 weeks
  Time to peak concentration (Tmax)
Pharmacokinetic characteristics. | 36 weeks
  Area under the drug concentration-time curve from time zero to the last measurable concentration time (AUC0-t)
Pharmacokinetic characteristics. | 36 weeks
  Elimination half-life (t1/2)
Pharmacokinetic characteristics. | 36 weeks
  Accumulation ratio based on AUC (Rac (AUC))
Pharmacokinetic characteristics. | 36 weeks
  Accumulation ratio based on peak concentration (Rac (Cmax))
Safety and tolerability | 36 weeks
  The incidence of AEs (adverse events) and SAEs (serious adverse events) from treatment until the last scheduled follow-up visit

SECONDARY OUTCOMES:
Changes from baseline in pre-bronchodilator FEV1 (forced expiratory volume at one second). | Weeks 0, 4, 8, 12, 24
  Changes in pre-bronchodilator FEV1 levels at 4, 8, 12, and 24 weeks compared to baseline.
Changes from baseline in post-bronchodilator FEV1. | Weeks 0, 4, 8, 12, 24
  Changes in post-bronchodilator FEV1 levels at 4, 8, 12, and 24 weeks compared to baseline.
Changes from baseline in post-brochodilator FEV1(%pred). | Weeks 0, 4, 8, 12, 24
  Changes in post-brochodilator FEV1(%pred) levels at 4, 8, 12, and 24 weeks compared to baseline.
Time to first moderate to severe Chronic Obstructive Pulmonary Disease Acute Exacerbation (AECOPD) from baseline to week 24. | Baseline to week 24.
  Time to first moderate to severe Chronic Obstructive Pulmonary Disease Acute Exacerbation (AECOPD) from baseline to week 24.
Annualized rate of moderate to severe AECOPD over the 24-week treatment period. | 24 weeks
Changes from baseline in mMRC(Modified Medical Research Council) dyspnea scale at 12 and 24 weeks. | Weeks 0, 12, 24
  Changes in mMRC dyspnea scale at 12 and 24 weeks compared to baseline.
Changes from baseline in CAT(COPD Assessment Test) score at 12 and 24 weeks. | Weeks 0, 12, 24
  Changes in CAT score at 12 and 24 weeks compared to baseline.
Incidence of ADAs Against 9MW1911. | 36 weeks
  The incidence of ADAs against 9MW1911 during the study will be summarized.

CONTACTS AND LOCATIONS:
Locations (22):
- China (22):
  - Baogang Hospital (No 3 Hospital Affiliated to Medical College of Inner Mongolia), Baotou
  - China-Japan Friendship Hospital, Beijing
  - Peking University Shougang Hospital, Beijing
  - The First Hospital of Changsha, Changsha
  - The second xiangya hospital of central south university, Changsha
  - Chengdu Fifth People's Hospital, Chengdu
  - Chongqing Red Cross Hospital (People's Hospital of Jiangbei District), Chongqing
  - Fu Yang People's Hospital, Fuyang
  - The First Affiliated Hospital of Guangzhou Medical University, Guangzhou
  - The Third Affiliated Hospital of Guangzhou Medical University, Guangzhou
  - The Second Hospital, University of South China, Hengyang
  - The Third People's Hospital of Huizhou, Huizhou
  - Jiangmen Central Hospital, Jiangmen
  - Liaocheng People's Hospital, Liaocheng
  - The First Affiliated Hospital of Nanchang University, Nanchang
  - Pingxiang People's Hospital, Pingxiang
  - The First Affiliated Hospital of Qiqihar Medical University, Qiqihar
  - Tongji Hospital of Tongji University, Shanghai
  - Shengjing Hospital of China Medical University, Shenyang
  - Suzhou Municipal Hospital, Suzhou
  - The First Hospital of Shanxi Medical University, Taiyuan
  - Taizhou Hospital of Zhejiang Province, Taizhou